CLINICAL TRIAL: NCT02783768
Title: Ventilation and Pulmonary Endothelium Toxicities (VaPE-Tox) of E-cigarettes: A Randomized Crossover Pilot Study
Brief Title: Ventilation and Pulmonary Endothelium Toxicities of E-cigarettes: A Randomized Crossover Pilot Study
Acronym: VaPE-Tox
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Elizabeth Oelsner, Assistant Professor of Medicine, Columbia University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: AAAQ8089
Record Dates: First submitted 2016-05-24; First posted 2016-05-26 (Estimated); Results first posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive; E-cigarettes
Keywords: E-cigarettes; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Vaping | interventions — salicylhydroxamic acid; Gadolinium

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- E-cigarette first (Experimental): Participants will undergo the e-cigarette exposure prior to the first two MRI measures, and then they will undergo the sham exposure prior to the last two MRI measures. The two MRIs performed under both experimental exposures (e-cigarette and sham) will be enhanced by (1) gadolinium and then (2) hyperpolarized 3-helium.
  Interventions: Device: E-cigarette; Other: Sham; Drug: Hyperpolarized 3-Helium; Drug: Gadolinium
- Sham first (Experimental): Participants will undergo the sham exposure prior to the first two MRI measures, and then they will undergo the e-cigarette exposure prior to the last two MRI measures. The two MRIs performed under both experimental exposures (e-cigarette and sham) will be enhanced by (1) gadolinium and then (2) hyperpolarized 3-helium.
  Interventions: Device: E-cigarette; Other: Sham; Drug: Hyperpolarized 3-Helium; Drug: Gadolinium

INTERVENTIONS:
Device: E-cigarette — The study e-cigarette exposure will be 10 puffs with 30-second inter-puff intervals, as directly observed by a trained research assistant, using a standardized e-cigarette. Cartomizers, batteries, and e-liquids will be obtained from commercial suppliers. The e-cigarette device will be loaded with 1 mL of flavorless e-liquid with a ratio of PG to vegetable glycerin of 70:30 and 1.8 mg/dL of nicotine.
Other: Sham — The "unexposed" condition will be breathing from the study e-cigarette (10 puffs with 30-second inter-puff intervals) with the battery off.
Drug: Hyperpolarized 3-Helium — Hyperpolarized 3-Helium will be used as an experimental contrast agent for the Ventilation MRIs performed twice per participant in both experimental arms. Approximately 250-600 mL of hyperpolarized 3He mixed with 300-750 mL nitrogen will be inhaled through a one-way valve in one inhalation starting approximately at residual volume.
  Other Names: 3-He
Drug: Gadolinium — Gadolinium contrast will be injected into the antecubital vein through an 18-20 gauge IV. The type of gadolinium will be 0.03 mmol/kg bodyweight of dotarem (gadoterate meglumine).
  Other Names: Gd

SUMMARY:
Determination of the acute pulmonary toxicities of e-cigarettes in young adults is of major public health importance, as e-cigarette vapor contains established toxicants that as hypothesized cause acute damage to the airways and the pulmonary microvasculature that may promote the development of CLD, for which there remain few effective therapies.

The study therefore propose a pilot study using a randomized crossover design in ten healthy young adults to test the acute effects of a standardized e-cigarette exposure on two sensitive, safe, non-invasive imaging measures: (1) ventilation defects on hyperpolarized helium-enhanced magnetic resonance imaging, and (2) pulmonary microvascular blood flow on gadolinium-enhanced pulmonary magnetic resonance angiography.

DETAILED DESCRIPTION:
Magnetic resonance imaging (MRI) and angiography (MRA) measures are promising approaches to detecting and characterizing the anticipated acute pulmonary toxicities of e-cigarettes. Hyperpolarized helium (3He)-enhanced MRI may be more sensitive than spirometry, a global lung function measure, for determination of airway toxicities. 3He-enhanced MRI has been used to demonstrate the extent of ventilation defects in healthy persons with normal spirometry; to measure ventilation changes in asthmatics pre- and post-challenge with bronchodilators and methacholine; and to predict pulmonary hospitalizations in persons with COPD. Meanwhile, until recently, non-invasive measures of pulmonary vascular toxicities were lacking. The investigators have developed an innovative measure of pulmonary microvascular blood flow on gadolinium (Gd)-enhanced MRA, which the investigators found to be markedly abnormal in early chronic obstructive pulmonary disease (COPD) and emphysema, and to be associated with increased endothelial microparticles, a marker of endothelial dysfunction. Nonetheless, neither of these sensitive, non-invasive, repeatable, and reproducible measures has ever been used to assess e-cigarette toxicities.

It is hypothesized that e-cigarette vapor inhalation will result in an acute increase in global and regional ventilation defects and an acute decrease in global and regional pulmonary microvascular perfusion.

This pilot work will provide the experience and data to support subsequent funding applications powered to definitively establish the acute toxicities of e-cigarette vapor of various compositions (e.g., with and without nicotine, with and without flavoring) in persons with and without chronic lung diseases (e.g., asthma) on pulmonary ventilation and microvascular perfusion. Furthermore, confirmation of the hypotheses in this sample would provide important preliminary evidence of e-cigarette pulmonary toxicities to inform interim regulatory decisions, as well as potentially generating vivid images of e-cigarette harms that may be meaningful to the general public and therefore suitable for use in public education campaigns.

ELIGIBILITY:
Inclusion Criteria:

* current use of e-cigarettes (>1x/month but <4 days/week)

Exclusion Criteria:

* any chronic medical or major psychiatric problems including current asthma
* self-reported heavy snoring/sleep apnea
* pre-bronchodilator FEV1 or FVC <80% predicted or FEV1/FVC < lower limit of normal
* MRI exclusions (pregnancy, claustrophobia, metal in body, gadolinium allergy, eGFR <60 mL/min/1.73m2)
* MRI scan with contrast within the last 12 months or planned MRI with contrast in the next 6 months
* use of any of the following in the prior 30 days: any conventional cigarettes, marijuana >10 days, any illicit drugs, any medication or inhalers (excluding hormonal contraceptives)
* binge drinking (≥5 alcoholic beverages over 2 hours) over the prior two weeks
* adverse symptomatic response to the study e-cigarette exposure (e.g., palpitations, shortness of breath, chest pain, headache, dizziness)

Ages: 21 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-07-24 (Actual); Study Completion 2018-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Oelsner, MD, MPH, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were a total of 12 subjects enrolled. 6 subjects were randomized to "E-cigarette first," of which 5 completed the full protocol. 5 subjects were randomized to "Sham first," all 5 of whom completed the full protocol. 1 subject was consented but not randomized.
Period: Overall Study
Arm/Group | E-cigarette First | Sham First
Started | 6 | 5
Completed | 5 | 5
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: There were a total of 12 subjects enrolled. 6 subjects were randomized to "E-cigarette first," of which 5 completed the full protocol. 5 subjects were randomized to "Sham first," all 5 of whom completed the full protocol. 1 subject was consented but not randomized and is therefore not included/reported in the baseline analysis population.
Groups:
- Total: This is a randomized crossover study. Participants were randomized to two groups, which differed by order of the exposure to e-cigarette versus sham: (1) e-cigarette first, followed by sham, or (2) sham first, followed by e-cigarette. All participants were both "exposed" and "unexposed."
Arm/Group | Total
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 1
  More than one race | 0
  Unknown or Not Reported | 6
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Pulmonary Microvascular Blood Flow (PMBF), Measured on Gadolinium-enhanced MRI, Between E-cigarette Exposed and Unexposed Conditions
Description: PMBF will be measured on gadolinium-enhanced MRI after e-cigarette and sham exposures. There were four days between the measurements of PMBF (e-cigarette) and PMBF (sham). PMBF is measured in mL(blood)/min/mL(lung volume). Lower PMBF has been observed in adults with COPD and emphysema.
Time Frame: After exposure (approximately 30 seconds)
Population: Since this study applied a randomized crossover design, participants from both randomization groups (exposure first and sham first) experienced both e-cigarette and sham exposures. In this outcome measure, the same 10 evaluable subjects all had exposure and no exposure at different time periods in the study.
Measure: Mean (Standard Deviation); unit: mL(blood)/min/mL(lung)
Groups:
- Exposed to E-cigarette: Participants were exposed to a standardized e-cigarette prior to MRI measurement of the outcome measure. Since this study applied a randomized crossover design, participants from both randomization groups (exposure first and sham first) are reported in this group.
- Unexposed (Sham): Participants were exposed to a standardized sham prior to MRI measurement of the outcome measure. Since this study applied a randomized crossover design, participants from both randomization groups (exposure first and sham first) are reported in this group.
Arm/Group | Exposed to E-cigarette | Unexposed (Sham)
Number analyzed (Participants) | 10 | 10
mL(blood)/min/mL(lung) | 74.4 (23.9) | 63.1 (19.4)
Statistical Analysis 1: Comparison: Exposed to E-cigarette vs Unexposed (Sham); Within-person effects of e-cigarette exposure on pulmonary microvascular blood flow (PMBF) was assessed via mixed models accounting for order effects. Null hypothesis: e-cigarette exposure is NOT associated with a change in PMBF. Alternative hypothesis: e-cigarette exposure IS associated with a change in PMBF. Power calculation: not applicable since this was a pilot/feasibility study; Test type: Other — Testing for difference in the outcome measure according to the exposure (which was not a treatment) in a randomized crossover setting; p = 0.012, Mixed Models Analysis; Mean Difference (Net) = 13.98, 95% CI 2-sided [4.012 to 23.94] — Measurements were included for participants with at least one valid MRI measurement

2. Primary Outcome: Ventilation Defect Percentage (VDP), Measured on Hyperpolarized 3-helium Enhanced MRI
Description: VDP will be measured on hyperpolarized 3Helium-enhanced MRI after e-cigarette and sham exposures. Due to limitations of prior qualitative/visual assessments of MRI, we developed and validated a new deep learning approach to the precise measurement of ventilation defects and report the percent non-fully ventilated lung using this method.
Time Frame: After exposure (approximately 30 seconds)
Population: A subset of participants were unable to complete the 3-He enhanced MRI due to problems with the helium polarizer and/or scanner (e.g., unable to fit into scanner due to body size). In this outcome measure, 7 out of 11 subjects had evaluable data.
Measure: Mean (Standard Deviation); unit: percentage of total lung volume
Arm/Group | Exposed to E-cigarette | Unexposed (Sham)
Number analyzed (Participants) | 7 | 7
percentage of total lung volume | 5.5 (4.4) | 6.6 (4.4)

3. Secondary Outcome: Regional PMBF, Measured on Gadolinium-enhanced MRI
Description: Regional PMBF (ie, in the right versus left, upper versus lower lobes) will be measured on gadolinium-enhanced MRI after e-cigarette and sham exposures.
Time Frame: After exposure (approximately 30 seconds)
Population: Data were not analyzed due to unavailable resources and technology because of the pandemic.
Arm/Group | Exposed to E-cigarette | Unexposed (Sham)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Regional VDP, Measured on Hyperpolarized 3-helium Enhanced MRI
Description: Regional VDP in the lower lung was measured on hyperpolarized 3Helium-enhanced MRI after e-cigarette and sham exposures.
Time Frame: After exposure (approximately 30 seconds)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of total lung volume
Arm/Group | Exposed to E-cigarette | Unexposed (Sham)
Number analyzed (Participants) | 7 | 7
percentage of total lung volume | 3.6 (2.8) | 5.8 (6.2)

5. Secondary Outcome: Lung Function, Measured on Spirometry
Description: Lung function will be measured on spirometry. Two participants had only one valid FEV1 measure, and one participant had no valid FEV1 measures. Hence, 3 participants (2 in "E-cigarette first" and 1 in "Sham first") were not analyzed. The analysis combines the groups in order to separate the effects of randomization group (order) and exposure.
Time Frame: After exposure (approximately 30 seconds)
Population: In this outcome measure, 7 out of 11 subjects had evaluable data.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Exposed to E-cigarette | Unexposed (Sham)
Number analyzed (Participants) | 7 | 7
L | 4.22 (0.75) | 4.08 (1.14)

6. Secondary Outcome: Diffusing Capacity of the Lung for Carbon Monoxide (DLCO)
Description: DLCO will be measured. There was a malfunction of the machine used to measure the DLCO. Hence, only one participant had paired DLCO values and 3 had unpaired measures.
Time Frame: After exposure (approximately 30 seconds)
Population: In this outcome measure, the machine broke and only 3 subjects had evaluable data for the exposed time period and 2 subjects had evaluable data for the unexposed time period
Measure: Mean (Standard Deviation); unit: mL/min/mm Hg
Arm/Group | Exposed to E-cigarette | Unexposed (Sham)
Number analyzed (Participants) | 3 | 2
mL/min/mm Hg | 33.65 (3.53) | 32.73 (8.69)

7. Secondary Outcome: Cardiac Output, Measured on Cardiac MRI
Description: Cardiac output will be measured on cardiac MRI. In the "E-cigarette first" arm, 2 participants did not have 2 valid measures of CO (one pair was missing, one was invalid). In the "Sham first" arm, 3 participants had one invalid measure of CO. The analysis combines the groups in order to separate the effects of randomization group (order) and exposure.
Time Frame: After exposure (approximately 30 seconds)
Population: In this outcome measure, 8 subjects had evaluable data for the exposed time period and 7 subjects had evaluable data for the unexposed time period.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Exposed to E-cigarette | Unexposed (Sham)
Number analyzed (Participants) | 8 | 7
mL/min | 6197 (1097) | 6093 (844)

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | E-cigarette First | Sham First
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 0/6 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-11): https://cdn.clinicaltrials.gov/large-docs/68/NCT02783768/Prot_SAP_000.pdf